CLINICAL TRIAL: NCT04734197
Title: A Multicenter, Randomized, Double-Masked Study To Evaluate The Safety, Tolerability, And Efficacy Of SURF-100 Ophthalmic Solution (A Mycophenolic Acid/Betamethasone Sodium Phosphate Combination) In Subjects With Dry Eye Disease
Brief Title: A Research Study To See How Well an Eye Drop, SURF-100 (A Mycophenolic Acid/Betamethasone Sodium Phosphate Combination), Works and What Side Effects There Are in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Surface Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-100-001
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Mycophenolic Acid; betamethasone sodium phosphate; Cyclosporine; Cyclosporins; lifitegrast; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- SURF-100 (a combination of 0.3% Mycophenolic Acid and 0.01% Betamethasone Sodium Phosphate) (Experimental): One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days
  Interventions: Drug: SURF-100 (Combination of 0.3% Mycophenolic Acid and 0.01% Betamethasone Sodium Phosphate)
- Mycophenolic Acid 0.1% (Experimental): One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
  Interventions: Drug: Mycophenolic Acid 0.1%
- Mycophenolic Acid 0.3% (Experimental): One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
  Interventions: Drug: Mycophenolic Acid 0.3%
- Betamethasone Sodium Phosphate 0.01% (Experimental): One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
  Interventions: Drug: Betamethasone Sodium Phosphate 0.01%
- Vehicle (Placebo Comparator): One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
  Interventions: Drug: Placebo Comparator: Vehicle
- Cyclosporine 0.05% Ophthalmic Emulsion (Active Comparator): One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days
  Interventions: Drug: Cyclosporine 0.05% Ophthalmic Emulsion
- Lifitegrast 5% Ophthalmic Solution (Active Comparator): One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days
  Interventions: Drug: Lifitegrast 5% Ophthalmic Solution

INTERVENTIONS:
Drug: SURF-100 (Combination of 0.3% Mycophenolic Acid and 0.01% Betamethasone Sodium Phosphate) — combination of a topical immunosuppressant and a topical corticosteroid solution
  Arms: SURF-100 (a combination of 0.3% Mycophenolic Acid and 0.01% Betamethasone Sodium Phosphate)
Drug: Mycophenolic Acid 0.1% — topical immunosuppressant
  Arms: Mycophenolic Acid 0.1%
Drug: Mycophenolic Acid 0.3% — topical immunosuppressant
  Arms: Mycophenolic Acid 0.3%
Drug: Betamethasone Sodium Phosphate 0.01% — topical corticosteroid solution
  Arms: Betamethasone Sodium Phosphate 0.01%
Drug: Placebo Comparator: Vehicle — topical vehicle solution
  Arms: Vehicle
Drug: Cyclosporine 0.05% Ophthalmic Emulsion — topical ophthalmic emulsion
  Other Names: Restasis 0.05% ophthalmic emulsion
  Arms: Cyclosporine 0.05% Ophthalmic Emulsion
Drug: Lifitegrast 5% Ophthalmic Solution — topical ophthalmic solution
  Other Names: Xiidra 5% Ophthalmic Solution
  Arms: Lifitegrast 5% Ophthalmic Solution

SUMMARY:
SURF-100 is being studied for the treatment of dry eye disease. SURF-100 is an investigational drug (which means the study drug is currently being tested) in the form of a sterile eye drop.

The purpose of this research study is to see how well SURF-100 works to treat dry eye and what potential side effects there are, and to compare it with Vehicle (placebo), 0.1% mycophenolic acid (MPA) in Vehicle, 0.3% MPA in Vehicle, 0.01% betamethasone phosphate (BSP) in Vehicle, Restasis and Xiidra. This study will involve about 280-350 study participants age 18 and older at about 40 different research sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 18 years of age at the time of the Screening visit.
2. Willing and able to read, sign, and date the informed consent form (ICF) after the nature of the study has been explained and any questions have been answered, and prior to initiation of any study procedures or exams.
3. Willing and able to comply with all study procedures and attend all study visits.
4. Willing to suspend use of tear substitutes at least 72 hours prior to Visit 2 (Day 0) through Visit 7 (Day 98).
5. Best corrected visual acuity (BCVA) of 0.7 log of the minimum angle of resolution (logMAR) or better (Snellen equivalent score of 20/100 or better) in each eye at Visit 1 (Day -14 to Day 0).
6. Subject-reported history of dry eye in both eyes.
7. Meeting ALL of the following criteria in the same eye at Visit 1 (Day -14 to Day 0) and meeting ALL of the following criteria in the same eye at Visit 2 (Day 0) if Visit 2 is performed >5 days after Visit 1:

   1. Minimum score of greater than or equal to 5 but less than or equal to 9 on UNC DEMS questionnaire.
   2. Schirmer Tear Test (with anesthesia) equal to or less than 10 mm, but more than 1 mm.
   3. TBUT: Equal to or less than 5 seconds
8. A negative urine pregnancy test if female and of childbearing potential (those who are not surgically sterilized [bilateral tubal ligation, hysterectomy, or bilateral oophorectomy] or post-menopausal [12 months after last menses] or premenarchal) and must have used adequate birth control throughout the study period (through Visit 7 [Day 98]). Adequate birth control is defined as hormonal-oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as condom or diaphragm; intrauterine device; abstinence; or surgical sterilization of male partner.
9. Subjects with secondary Sjögren's syndrome (e.g., rheumatoid arthritis, systemic lupus erythematosus) or other autoimmune diseases (e.g., multiple sclerosis, inflammatory bowel disease) are eligible for study consideration provided the subject meets all other inclusion and exclusion criteria, AND are not in a medical state - in the opinion of the principal investigator - that could interfere with study parameters, are not taking systemic/ocular steroids, and are not immunodeficient/immunosuppressed (e.g., receiving systemic immunomodulating or immunosuppressive drugs to manage their baseline medical state).

Exclusion Criteria:

1. Contraindications or known hypersensitivity to the study drug(s), including RESTASIS or XIIDRA, or their components.
2. Subjects who are employees or immediate family members of employees at the investigational site.
3. Subjects who are members of the same household.
4. Any ocular condition that, in the opinion of the investigator, may affect study parameters including, but not limited to, lid margin disorders (e.g., blepharitis including staphylococcal, demodex, or seborrheic; excessive lid laxity, floppy eyelid syndrome, ectropion, entropion), advanced conjunctivochalasis, Salzmann's nodular degeneration, and asthenopia-related conditions, allergic conjunctivitis, glaucoma, diabetic retinopathy, follicular conjunctivitis, iritis, uveitis, wet-exudative age-related macular degeneration, retinal vein occlusion, and/or active ocular inflammation.
5. Any condition that could affect trigeminal nerve function including facial or ocular Herpes Zoster/Shingle, a stroke or nerve palsy affecting the eye(s).
6. Use of any topical medication and/or antibiotics for the treatment of blepharitis or meibomian gland disease in either eye within 14 days prior to Visit 2 (Day 0).
7. Active or history of ocular herpes or any other ocular infection in either eye within the last 30 days prior to Visit 1 (Day -14 to Day 0).
8. Unwilling to avoid wearing contact lenses for 7 days prior to Randomization (Visit 2, Day 0) and for the duration of the study period (through Visit 7, Day 98).
9. Positive urine pregnancy test at Screening, nursing an infant or planning to become pregnant during the study.
10. Any blood donation or significant loss of blood within 56 days of Visit 1 (Day -14 to Day 0).
11. Any history of immunodeficiency disorder, human immunodeficiency virus (HIV), positive hepatitis B, C, or evidence of acute active hepatitis A (anti-hepatitis A virus immunoglobulin M), or organ or bone marrow transplant.
12. Any medication (oral or topical) known to cause ocular drying that is not administered as a stable dose for at least 30 days prior to Visit 1 (Day -14 to Day 0) and for the duration of the study (Visit 7, Day 98); antihistamines are not allowed at any time during the study.
13. Use of prohibited medications (topical, topical ophthalmic and/or systemic, during the appropriate pre-study washout period (see below) and during the study. Prohibited medications include topical cyclosporine or lifitegrast, use of any other ophthalmic medication (e.g., glaucoma medication, topical anti-inflammatory eye drops) for the duration of the study)

    NOTE: Supplements containing omega-3 are allowed if the subject has been taking said supplement for at least 3 months prior to Screening. Subjects are not allowed to begin taking supplements containing omega-3 during the study. The appropriate pre-study washout period is as follows:
    1. Antihistamines (including ocular): 7 days prior to Visit 1 (Day -14 to Day 0).
    2. Topical cyclosporine or lifitegrast or omega-3s within 14 days prior to Visit 1 (Day -14 to Day 0).
    3. Corticosteroids or mast cell stabilizers (including ocular): 14 days prior to Visit 1 (Day -14 to Day 0).
    4. Depot-corticosteroids in either eye at least 45 days prior to the first dose of study drug (Day 0)
    5. All other topical ophthalmic preparations (including artificial tear substitutes other than the study drops): 72 hours prior to Visit 1 (Day -14 to Day 0).
    6. Introduction of any new, nonsteroidal anti-inflammatory drugs (NSAIDs) including but not limited to topical, systemic (including sleep-aids containing NSAIDs), inhaled, or irrigation solution within 7 days prior to the first dose of study drug. Subjects who are on stable dose of NSAIDs (stable for at least 4 weeks prior to the first dose of study drug) are eligible for participation and should remain on a stable dose throughout the duration of the study (i.e., through Day 98).
    7. Triamcinolone in either eye at least 90 days prior to the first dose of study drug (Day 0).
    8. Inhaled, ingested, sublingual, transdermal or topical products containing marijuana, tetrahydrocannabinol (THC) or cannabidiol (CBD) at least 7 days prior to the first dose of study drug (Day 0).
    9. Systemic pain relievers, analgesics (e.g., pregabalin, gabapentin, opioids) 14 days prior to the first dose of study drug (Day 0).
    10. Any supplement, prescribed medication or over-the-counter product that the investigator feels may interfere with the study parameters, including homeopathic remedies, analgesics, and pain medication.
    11. Oral doxycycline within 6 months of first dose of study drug (Day 0).
    12. Diuretics: Within 28 days prior to Visit 1 (Day -14 to Day -1).
    13. Punctal occlusion:

    i. Punctal cauterization: Randomization may not occur until 4 weeks following the procedure.

    ii. Permanent/semi-permanent punctal plugs (this includes 180-day punctal plugs): Randomization may not occur until 4 weeks following the procedure. If a punctal plug falls out during the study, it should be reinserted.

    iii. Temporary collagen punctal plugs: Not permitted. If subject has a history of use of temporary punctal plugs, randomization may not occur until 4 weeks since last insertion and puncta are plug-free, as determined by the investigator.
14. Any significant chronic illness that, in the opinion of the investigator, could interfere with the study parameters, including, but not limited to, severe cardiopulmonary disease, poorly controlled hypertension, and/or poorly controlled diabetes.
15. Use of any investigational product or device within 30 days prior to Visit 1 (Day -14 to Day 0) or during the study period.
16. History of LASIK or similar type of corneal refractive surgery within 12 months prior to Visit 1 (Day -14 to Day 0), and/or any other ocular surgical procedure within 12 months prior to Visit 1 (Day -14 to Day 0); or any scheduled ocular surgical procedure during the study period.
17. Use of any laser procedure for the eyes in the 30 days prior to Visit 1 (Day -14 to Day 0).
18. Known history of alcohol and/or drug abuse within the past 12 months that in the opinion of the principal investigator, may interfere with study compliance, outcome measures including safety parameters, and/or the general medical condition of the subject.
19. Subjects with dry eye secondary to scarring (such as that seen with irradiation, alkali burns, Stevens Johnson syndrome, cicatricial pemphigoid) or destruction of conjunctival goblet cells (as with vitamin A deficiency) are not eligible for the study. Subjects with incidental scars secondary to refractory surgery (i.e., LASIK surgery) that, in the opinion of the principal investigator, would not interfere with study compliance and/or outcome measures, are not excluded from the study.
20. Subjects who test positive for the COVID-19 virus within 30 days prior to Visit 1 (Day -14 to Day 0).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Hosseini, MD, PhD, Study Chair — Surface Ophthalmics, Inc. (formerly Surface Pharmaceutials, Inc.)
Locations (40):
- United States (40):
  - Cornea and Cataract Consultants of Arizona PC, Phoenix, Arizona
  - Canyon City EyeCare, Azusa, California
  - Inland Eye Specialists, Hemet, California
  - North Valley Eye Medical Group Inc., Mission Hills, California
  - LoBue Laser and Eye Medical Center, Murrieta, California
  - Eye Research Foundation, Newport Beach, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Sacramento Eye Consultants, A Medical Corporation, Sacramento, California
  - The Eye Center of Northern Colorado, Fort Collins, Colorado
  - Connecticut Eye Consultants, PC, Danbury, Connecticut
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - Hernando Eye Institute, Brooksville, Florida
  - Bowden Eye and Associates, Jacksonville, Florida
  - Eye Center of North Florida PA, Panama City, Florida
  - International Research Center, Tampa, Florida
  - Blue Ocean Clinical Research at The Macula Center, The Villages, Florida
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Jackson Eye, Lake Villa, Illinois
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Kentucky Eye Institute, Lexington, Kentucky
  - Midwest Vision Research Foundation at Pepose Vision Institute, Chesterfield, Missouri
  - Tauber Eye Center, Kansas City, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Ophthalmology Consultants Ltd., St Louis, Missouri
  - EyeSight Ophthalmic Services, Somersworth, New Hampshire
  - Alterman, Modi & Wolter, Poughkeepsie, New York
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Physicians Protocol, Greensboro, North Carolina
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Total Eye Care, PA, Memphis, Tennessee
  - VRF Eye Specialty Group, Memphis, Tennessee
  - West TN EyeCare dba Toyos Clinic, Nashville, Tennessee
  - Texan Eye Care, PA - Keystone Research, Ltd, Austin, Texas
  - Houston Eye Associates, Houston, Texas
  - Advanced Laser Vision & Surgical Institute, Houston, Texas
  - Eye Clinics of South Texas, PA, San Antonio, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - Tanner Clinic, Layton, Utah
  - The Eye Institute of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to each participant's assignment by chance to one of the seven treatment arms/groups (randomization), the Investigator designated the participant's Study Eye. The participant's Study Eye was the eye that was eligible for the study and had the worst signs and symptoms. The participant's other eye was called the Fellow Eye.
Units Other Than Participants: Study Eyes
Groups:
- SURF-100: Eye drop:
  Topical, preservative-free SURF-100 (a combination of 0.3% mycophenolic acid and 0.01% betamethasone sodium phosphate)
  Dosing: One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
- Mycophenolic Acid 0.1%: Eye drop:
  Topical, preservative-free mycophenolic acid 0.1%
  Dosing: One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
- Mycophenolic Acid 0.3%: Eye drop:
  Topical preservative-free mycophenolic acid 0.3%
  Dosing: One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
- Betamethasone Sodium Phosphate 0.01%: Eye drop:
  Topical preservative free betamethasone sodium phosphate 0.01%
  Dosing: One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
- Placebo Comparator: Vehicle: Eye drop:
  Topical preservative-free placebo comparator (vehicle)
  Dosing: One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
- Cyclosporine 0.05% Ophthalmic Emulsion: Eye drop:
  Topical preservative-free cyclosporine 0.05% ophthalmic emulsion
  Dosing: One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
- Lifitegrast 5% Ophthalmic Solution: Eye drop:
  Topical, preservative-free lifitegrast 5% ophthalmic solution
  Dosing: One drop in the study eye (and fellow eye, if applicable) twice daily for 84 days.
Period: Overall Study
Arm/Group | SURF-100 | Mycophenolic Acid 0.1% | Mycophenolic Acid 0.3% | Betamethasone Sodium Phosphate 0.01% | Placebo Comparator: Vehicle | Cyclosporine 0.05% Ophthalmic Emulsion | Lifitegrast 5% Ophthalmic Solution
Started | 52; 52 Study Eyes | 50; 50 Study Eyes | 50; 50 Study Eyes | 49; 49 Study Eyes | 47; 47 Study Eyes | 47; 47 Study Eyes | 54; 54 Study Eyes
Completed | 44; 44 Study Eyes | 46; 46 Study Eyes | 44; 44 Study Eyes | 44; 44 Study Eyes | 44; 44 Study Eyes | 43; 43 Study Eyes | 43; 43 Study Eyes
Not Completed | 8; 8 Study Eyes | 4; 4 Study Eyes | 6; 6 Study Eyes | 5; 5 Study Eyes | 3; 3 Study Eyes | 4; 4 Study Eyes | 11; 11 Study Eyes

BASELINE CHARACTERISTICS:
Population: All subjects randomized are included.
Units Other Than Participants: Study Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | SURF-100 | Mycophenolic Acid 0.1% | Mycophenolic Acid 0.3% | Betamethasone Sodium Phosphate 0.01% | Placebo Comparator: Vehicle | Cyclosporine 0.05% Ophthalmic Emulsion | Lifitegrast 5% Ophthalmic Solution | Total
Number analyzed (Participants) | 52 | 50 | 50 | 49 | 47 | 47 | 54 | 349
Number analyzed (Study Eyes) | 52 | 50 | 50 | 49 | 47 | 47 | 54 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (14.16) | 61.4 (16.29) | 60.3 (14.34) | 61.8 (13.92) | 60.7 (14.75) | 63.2 (13.41) | 62.8 (14.53) | 61.7 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 39 | 44 | 35 | 34 | 41 | 265
  Male | 15 | 15 | 11 | 5 | 12 | 13 | 13 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 4 | 1 | 1 | 4 | 3 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 2 | 1 | 6 | 2 | 7 | 6 | 31
  White | 40 | 42 | 47 | 41 | 41 | 36 | 44 | 291
  More than one race | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 6
University of North Carolina Dry Eye Management Scale (UNC DEMS) Score at Baseline [Mean (Standard Deviation); unit: UNC DEMS units] — The UNC DEMS scale is a participant-specific 10-point scale with a minimum score of 1 ([1-2] My symptoms are not a problem. My dry eye does not affect my daily life at all) and a maximum score of 10 ([9-10] my symptoms are severe and I need immediate medical care. My dry eye greatly affects my daily life).
  UNC DEMS units | 7.1 (1.13) | 6.9 (1.23) | 6.7 (1.33) | 6.7 (1.11) | 7.0 (1.19) | 6.8 (1.07) | 6.9 (1.32) | 6.9 (1.20)
Tear Break-up Time (TBUT), Study Eye [Mean (Standard Deviation); unit: seconds] — Tear break-up time (TBUT) is a method used to assess the stability of tear film. TBUT is the time it takes for the first dry spot to appear on the cornea after a complete blink.
  seconds | 3.43 (0.98) | 3.60 (0.87) | 3.41 (0.91) | 3.39 (0.87) | 3.62 (0.83) | 3.36 (0.78) | 3.43 (0.88) | 3.5 (0.88)
Schirmer Tear Test (with Anesthesia), Study Eye [Mean (Standard Deviation); unit: millimeters] — The Schirmer test is a method to assess whether the eye produces enough tears to keep it moist. In this study it was performed with anesthesia.
  millimeters | 5.7 (2.48) | 5.1 (2.42) | 5.2 (2.54) | 5.8 (2.70) | 5.6 (2.34) | 5.4 (2.48) | 5.5 (2.38) | 5.5 (2.47)

OUTCOME MEASURES:

1. Primary Outcome: University of North Carolina Dry Eye Management Scale (UNC DEMS) Responder Analysis
Description: The UNC DEMS scale is a participant-specific 10-point scale with a minimum score of 1 ([1-2] My symptoms are not a problem. My dry eye does not affect my daily life at all) and a maximum score of 10 ([9-10] my symptoms are severe and I need immediate medical care. My dry eye greatly affects my daily life).
  Participants with a 10% or higher reduction in UNC DEMS score from baseline were defined as responders, and response rates were summarized by treatment group.
Time Frame: Baseline and Day 84
Population: Intent-to Treat Analysis Population: Includes all randomized subjects. Missing values were imputed using last observation carried forward (LOCF).
  LOCF: common statistical approach to the analysis of longitudinal repeated measures where some follow-up [FU] observations may be missing.
  In a LOCF analysis, a missing FU value is replaced by/imputed as that participant's previously observed value. The combination of the observed and imputed data is then analyzed as if there were no missing data.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | SURF-100 | Mycophenolic Acid 0.1% | Mycophenolic Acid 0.3% | Betamethasone Sodium Phosphate 0.01% | Placebo Comparator: Vehicle | Cyclosporine 0.05% Ophthalmic Emulsion | Lifitegrast 5% Ophthalmic Solution
Number analyzed (Participants) | 52 | 50 | 50 | 49 | 47 | 47 | 54
percentage of responders | 65.4 [50.9 to 78.0] | 90.0 [78.2 to 96.7] | 66.0 [51.2 to 78.8] | 71.4 [56.7 to 83.4] | 80.9 [66.7 to 90.9] | 72.3 [57.4 to 84.4] | 57.4 [43.2 to 70.8]
Statistical Analysis 1: Comparison: SURF-100 vs Mycophenolic Acid 0.1% vs Mycophenolic Acid 0.3% vs Betamethasone Sodium Phosphate 0.01% vs Placebo Comparator: Vehicle vs Cyclosporine 0.05% Ophthalmic Emulsion vs Lifitegrast 5% Ophthalmic Solution; Exploratory Phase 2 Study; the sample size of approximately 280-350 subjects (between 40 and 50 subjects per each of the 7 treatment groups) was based on medical judgement; Test type: Superiority; p = 0.0040, Fisher Exact — The threshold for statistical significance is p=0.05

2. Secondary Outcome: Tear Break Up Time (TBUT), Study Eye
Description: The absolute change from baseline in TBUT in the study eye at Day 84.
Time Frame: Baseline and Day 84
Population: Intent-to Treat Analysis Population: It included all randomized subjects regardless of whether a study medication was taken. Missing data were not imputed. For subjects who were withdrawn from the study prior to study completion, all data compiled up to the point of subject withdrawal from the study was used for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Units Other Than Participants: Study Eyes
Arm/Group | SURF-100 | Mycophenolic Acid 0.1% | Mycophenolic Acid 0.3% | Betamethasone Sodium Phosphate 0.01% | Placebo Comparator: Vehicle | Cyclosporine 0.05% Ophthalmic Emulsion | Lifitegrast 5% Ophthalmic Solution
Number analyzed (Participants) | 50 | 50 | 50 | 49 | 47 | 47 | 52
Number analyzed (Study Eyes) | 50 | 50 | 50 | 49 | 47 | 47 | 52
seconds | 1.70 [0.52 to 2.88] | 1.84 [0.68 to 3.00] | 1.41 [0.21 to 2.60] | 2.56 [1.38 to 3.75] | 1.12 [-0.08 to 2.33] | 2.40 [1.20 to 3.59] | 1.52 [0.37 to 2.68]
Statistical Analysis 1: Comparison: SURF-100 vs Mycophenolic Acid 0.1% vs Mycophenolic Acid 0.3% vs Betamethasone Sodium Phosphate 0.01% vs Placebo Comparator: Vehicle vs Cyclosporine 0.05% Ophthalmic Emulsion vs Lifitegrast 5% Ophthalmic Solution; Mixed Model for Repeated Measures (MMRM) analysis included fixed effects of baseline TBUT, age, treatment, visit, and treatment by visit interaction. Least squares means (LSMs) of the absolute TBUT change from baseline and their 95% CIs were estimated from the MMRM model for each treatment group; Test type: Superiority; p = 0.3111, Fisher Exact; The threshold for statistical significance is p=0.05

3. Secondary Outcome: Schirmer Tear Test Score, Study Eye
Description: The absolute change from baseline in Schirmer tear score in the study eye at Day 84.
Time Frame: Baseline and Day 84
Population: Intent-to Treat (ITT) Analysis Population: It included all randomized subjects regardless of whether a study medication was taken. Missing data were not imputed. For subjects who were withdrawn from the study prior to study completion, all data compiled up to the point of subject withdrawal from the study was used for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Units Other Than Participants: Study Eyes
Arm/Group | SURF-100 | Mycophenolic Acid 0.1% | Mycophenolic Acid 0.3% | Betamethasone Sodium Phosphate 0.01% | Placebo Comparator: Vehicle | Cyclosporine 0.05% Ophthalmic Emulsion | Lifitegrast 5% Ophthalmic Solution
Number analyzed (Participants) | 50 | 50 | 50 | 49 | 47 | 47 | 52
Number analyzed (Study Eyes) | 50 | 50 | 50 | 49 | 47 | 47 | 52
millimeters | 3.20 [1.52 to 4.88] | 2.94 [1.32 to 4.57] | 4.46 [2.77 to 6.15] | 1.66 [0.00 to 3.33] | 3.98 [2.29 to 5.66] | 2.25 [0.57 to 3.92] | 2.73 [1.10 to 4.35]
Statistical Analysis 1: Comparison: SURF-100 vs Mycophenolic Acid 0.1% vs Mycophenolic Acid 0.3% vs Betamethasone Sodium Phosphate 0.01% vs Placebo Comparator: Vehicle vs Cyclosporine 0.05% Ophthalmic Emulsion vs Lifitegrast 5% Ophthalmic Solution; MMRM analysis included fixed effects of baseline Schirmer test score, age, treatment, visit, and treatment by visit interaction. LSMs of the absolute change from baseline in Schirmer test score and their 95% CIs were estimated from the MMRM model for each treatment group; Test type: Superiority; p = 0.2027, Fisher Exact — The threshold for statistical significance is p=0.05

ADVERSE EVENTS:
Time Frame: From each participant's signature of informed consent at Screening through Day 98 (completion of the study) or early withdrawal, which ever came first.
Description: Adverse events were collected from each participant's signature of informed consent at Screening through Day 98 (completion of the study) or early withdrawal, which ever came first.
Arm/Group | SURF-100 | Mycophenolic Acid 0.1% | Mycophenolic Acid 0.3% | Betamethasone Sodium Phosphate 0.01% | Placebo Comparator: Vehicle | Cyclosporine 0.05% Ophthalmic Emulsion | Lifitegrast 5% Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50 | 0/50 | 0/49 | 0/47 | 0/47 | 0/54
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/50 | 1/50 | 0/49 | 0/47 | 1/47 | 0/54
Other Adverse Events (participants affected / at risk) | 10/52 | 10/50 | 9/50 | 3/49 | 6/47 | 6/47 | 20/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SURF-100 (N=52) | Mycophenolic Acid 0.1% (N=50) | Mycophenolic Acid 0.3% (N=50) | Betamethasone Sodium Phosphate 0.01% (N=49) | Placebo Comparator: Vehicle (N=47) | Cyclosporine 0.05% Ophthalmic Emulsion (N=47) | Lifitegrast 5% Ophthalmic Solution (N=54)
Ocular hypertension not related to study drug (pre-existing condition) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Pre-existing condition - the study protocol required to report "an IOP of 30 mmHg or higher" as serious adverse event (SAE). The elevated IOP at screening was reported as a mild, non-treatment emergent SAE of ocular hypertension in both eyes.
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Moderate non-ocular treatment-emergent SAE that was considered by the Investigator to be unrelated to the study drug.
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Severe non-ocular treatment-emergent SAE that was considered by the Investigator to be unrelated to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SURF-100 (N=52) | Mycophenolic Acid 0.1% (N=50) | Mycophenolic Acid 0.3% (N=50) | Betamethasone Sodium Phosphate 0.01% (N=49) | Placebo Comparator: Vehicle (N=47) | Cyclosporine 0.05% Ophthalmic Emulsion (N=47) | Lifitegrast 5% Ophthalmic Solution (N=54)
Conjuctival hyperaemia, study eye and/or fellow eye (Eye disorders) | 3 (4) | 7 (8) | 4 (6) | 3 (4) | 6 (9) | 3 (4) | 0 (0)
Vision blurred, study eye and/or fellow eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (12)
Instillation site pain, study eye and/or fellow eye (General disorders) | 7 (11) | 3 (4) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 10 (10)
Instillation site pruritus, study eye and/or fellow eye (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT04734197/Prot_SAP_000.pdf